CLINICAL TRIAL: NCT01384552
Title: Do Weight Status and the Level of Dietary Restraint Moderate the Relationship Between Package Unit Size and Food Intake?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 8573 B
Record Dates: First submitted 2011-06-25; First posted 2011-06-29 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Overweight
Keywords: normal weight; overweight; dietary restraint; package unit size; food intake
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Normal Weight, Unrestrained - Standard (Active Comparator): Each participant is of normal weight (BMI: 18.5-24.9 kg/m2) and is classified as an unrestrained eater (scoring less than or equal to 12 on the Three Factor Eating Questionnaire - Cognitive Restraint Scale).
  Interventions: Other: Package Unit Size - Standard
- Normal Weight, Restrained - Single Serving (Active Comparator): Each participant is of normal weight (BMI: 18.5-24.9 kg/m2) and is classified as a restrained eater (scoring greater than 12 on the Three Factor Eating Questionnaire - Cognitive Restraint Scale).
  Interventions: Other: Package Unit Size - Single Serving
- Normal Weight, Restrained - Standard (Active Comparator): Each participant is of normal weight (BMI: 18.5-24.9 kg/m2) and is classified as a restrained eater (scoring greater than 12 on the Three Factor Eating Questionnaire - Cognitive Restraint Scale).
  Interventions: Other: Package Unit Size - Standard
- Overweight, Unrestrained - Single Serving (Active Comparator): Each participant is overweight (BMI: 25-39.9 kg/m2) and is classified as an unrestrained eater (scoring less than or equal to 12 on the Three Factor Eating Questionnaire - Cognitive Restraint Scale).
  Interventions: Other: Package Unit Size - Single Serving
- Overweight, Unrestrained - Standard (Active Comparator): Each participant is overweight (BMI: 25-39.9 kg/m2) and is classified as an unrestrained eater (scoring less than or equal to 12 on the Three Factor Eating Questionnaire - Cognitive Restraint Scale).
  Interventions: Other: Package Unit Size - Standard
- Overweight, Restrained - Single Serving (Active Comparator): Each participant is overweight (BMI: 25-39.9 kg/m2) and is classified as a restrained eater (scoring greater than 12 on the Three Factor Eating Questionnaire - Cognitive Restraint Scale).
  Interventions: Other: Package Unit Size - Single Serving
- Overweight, Restrained - Standard (Active Comparator): Each participant is overweight (BMI: 25-39.9 kg/m2) and is classified as a restrained eater (scoring greater than 12 on the Three Factor Eating Questionnaire - Cognitive Restraint Scale).
  Interventions: Other: Package Unit Size - Standard
- Normal Weight, Unrestrained - Single Serving (Active Comparator): Each participant is of normal weight (BMI: 18.5-24.9 kg/m2) and is classified as an unrestrained eater (scoring less than or equal to 12 on the Three Factor Eating Questionnaire - Cognitive Restraint Scale).
  Interventions: Other: Package Unit Size - Single Serving

INTERVENTIONS:
Other: Package Unit Size - Single Serving — Participants will receive a box of twenty-two, 0.9-oz. packages of pretzels. Participants will receive the box of pretzels in the lab on a Thursday or Friday and will take the box of pretzels home for a period of four days. Participants will bring back the box of pretzels to the lab on the following Monday or Tuesday (depending on the day of the initial receipt of pretzels).
  Arms: Normal Weight, Restrained - Single Serving; Normal Weight, Unrestrained - Single Serving; Overweight, Restrained - Single Serving; Overweight, Unrestrained - Single Serving
Other: Package Unit Size - Standard — Participants will receive a box of two, 10-oz. packages of pretzels. Participants will receive the box of pretzels in the lab on a Thursday or Friday and will take the box of pretzels home for a period of four days. Participants will bring back the box of pretzels to the lab on the following Monday or Tuesday (depending on the day of the initial receipt of pretzels).
  Arms: Normal Weight, Restrained - Standard; Normal Weight, Unrestrained - Standard; Overweight, Restrained - Standard; Overweight, Unrestrained - Standard

SUMMARY:
The objective of this study is to determine the independent and combined effects of weight status and the level of dietary restraint on the relationship between package unit size and food intake.

DETAILED DESCRIPTION:
The estimated prevalence of obesity among adults in 2007-2008 was 33.8% and the combined estimated prevalence of overweight and obesity was 68.0% [1]. Although there are no clear reasons for the current obesity epidemic, there is a general consensus that environmental dietary factors, such as package unit size, encourage excessive food intake and positive energy balance [2, 3]. It is believed that the package unit size of food indirectly influences food intake by impacting the accuracy of consumption monitoring [2, 4]. Large packages decrease the accuracy of consumption monitoring by making it difficult to assess how many servings have been consumed in one sitting, while small single-serving packages can increase the accuracy of consumption monitoring by providing a clear definition of what a standard serving is and how much one has consumed [2, 4, 5]. Therefore, it has been proposed that small, single-serving packages of snack foods may help reduce energy intake [4, 5]. To date, limited studies have been conducted in this area and the results are inconsistent [4-9]. Mixed results could be related to differences in participant variables, specifically weight status and level of dietary restraint (a term that refers to the amount of control exerted over food intake) [4, 9]. These individual characteristics may interact with food package unit size to influence one's food intake [2, 4]. Overweight individuals or restrained eaters may more closely monitor the volume of food they consume as compared to normal weight or unrestrained eaters [4, 9]. The [smaller] size of food packaging may aid in monitoring food consumption and thus, influence how much food is consumed in overweight and/or restrained eaters [2, 4]. Therefore, the objective of this study is to determine if weight status and the level of dietary restraint moderate the relationship between package unit size and food intake.

Specific Aims:

1. Determine the effect of dietary restraint on the relationship between package unit size and food intake.
2. Determine the effect of weight status on the relationship between package unit size and food intake.
3. Determine the combined effect of weight status and dietary restraint on the relationship between package unit size and food intake.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged 18-35 years old.
* Body Mass Index (BMI) between 18.5-24.9 kg/m2 or BMI between 25-39.9 kg/m2.

  * For normal weight groups: BMI of 18.5-24.9 kg/m2.
  * For overweight groups: BMI of 25-39.9 kg/m2.
* Dietary restraint scores of either less than or equal to 12 or > 12 on the Three Factor Eating Questionnaire-Cognitive Restraint scale (TFEQ-R) [10].

  * For unrestrained groups: less than or equal to 12.
  * For restrained groups: > 12.
* Do not have unfavorable preference toward pretzels.
* Do not have allergies to pretzel ingredients.
* Do not have a health condition or use medication that affects eating or requires a therapeutic diet.
* Must have a consistent schedule during the time of the study.
* Must agree to instructions to not share pretzel snack packages with others.

Exclusion Criteria:

* BMI below 18.5 or above 39.9 kg/m2.
* Have an unfavorable preference toward pretzels.
* Have allergies to pretzel ingredients (wheat flour).

  * Severe allergies to nuts - Synder's of Hanover pretzels are made in a facility that handles peanut butter.
* Are unwilling to consume pretzels during the time of the study.
* Are pregnant or breastfeeding.
* Do not meet one or more of the other above mentioned eligibility requirements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Total grams of pretzels consumed. | 4 days
  Total grams of pretzels consumed by participants over the 4-day study period will be determined by subtracting pre- and post-consumption weight of snack packages provided.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, Ph.D., Principal Investigator — University of Tennessee, Knoxville; Chrystal L Haire, B.S., Principal Investigator — University of Tennessee, Knoxville
Locations (1):
- Healthy Eating and Activity Laboratory, Knoxville, Tennessee, United States

REFERENCES:
- [Background] Flegal KM, Carroll MD, Ogden CL, Curtin LR. Prevalence and trends in obesity among US adults, 1999-2008. JAMA. 2010 Jan 20;303(3):235-41. doi: 10.1001/jama.2009.2014. Epub 2010 Jan 13. PMID 20071471
- [Background] French SA, Story M, Jeffery RW. Environmental influences on eating and physical activity. Annu Rev Public Health. 2001;22:309-35. doi: 10.1146/annurev.publhealth.22.1.309. PMID 11274524
- [Background] Wansink B. Environmental factors that increase the food intake and consumption volume of unknowing consumers. Annu Rev Nutr. 2004;24:455-79. doi: 10.1146/annurev.nutr.24.012003.132140. PMID 15189128
- [Background] Raynor HA, Wing RR. Package unit size and amount of food: do both influence intake? Obesity (Silver Spring). 2007 Sep;15(9):2311-9. doi: 10.1038/oby.2007.274. PMID 17890500
- [Background] Stroebele N, Ogden LG, Hill JO. Do calorie-controlled portion sizes of snacks reduce energy intake? Appetite. 2009 Jun;52(3):793-796. doi: 10.1016/j.appet.2009.02.015. Epub 2009 Mar 6. PMID 19501784
- [Background] Devitt AA, Mattes RD. Effects of food unit size and energy density on intake in humans. Appetite. 2004 Apr;42(2):213-20. doi: 10.1016/j.appet.2003.10.003. PMID 15010185
- [Background] Raynor HA, Van Walleghen EL, Niemeier H, Butryn ML, Wing RR. Do food provisions packaged in single-servings reduce energy intake at breakfast during a brief behavioral weight-loss intervention? J Am Diet Assoc. 2009 Nov;109(11):1922-5. doi: 10.1016/j.jada.2009.08.009. PMID 19857636
- [Background] Freedman MR, Brochado C. Reducing portion size reduces food intake and plate waste. Obesity (Silver Spring). 2010 Sep;18(9):1864-6. doi: 10.1038/oby.2009.480. Epub 2009 Dec 24. PMID 20035274
- [Background] Wansink B, Payne CR, Shimizu M. The 100-calorie semi-solution: sub-packaging most reduces intake among the heaviest. Obesity (Silver Spring). 2011 May;19(5):1098-100. doi: 10.1038/oby.2010.306. Epub 2011 Jan 13. PMID 21233814
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- See also: This is the website for the Healthy Eating and Activity Laboratory (HEAL), where this study is being conducted. — http://heal.utk.edu/